CLINICAL TRIAL: NCT06755710
Title: Patient Engagement in PTSD Treatment (PEP) - Advancing PTSD Treatment Outcomes
Brief Title: Patient Engagement in PTSD Treatment (PEP)
Acronym: PEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Anna Bolette Lund Nielsen, MD, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24049563
Record Dates: First submitted 2024-12-13; First posted 2025-01-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-12

CONDITIONS: PTSD; Depression Disorders; Patient Engagement
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Patient Participation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment as usual (TAU) (Active Comparator): 8-12 months of treatment Interventions: Behavioral: treamtent as usuan (TAU)
  Interventions: Behavioral: Treatment as Usual
- Introductory PTSD module + TAU (Experimental): 9-13 months of treatment An intervention with an introductory PTSD module consistent of four sessions focusing on motivation followed by TAU
  Interventions: Behavioral: Introductory PTSD module; Behavioral: Treatment as Usual
- Introductory PTSD module + one session of Shared Decision Making + individualised treatment (Experimental): 9-13 months of treatment Add-on introductory PTSD module and add-on patient-centred shared decision making session before continuing in the chosen standardised treatment.
  Interventions: Behavioral: Introductory PTSD module; Behavioral: Shared Decision Making; Behavioral: Standardised treatments

INTERVENTIONS:
Behavioral: Introductory PTSD module — The Introductory PTSD module consist of four session focusing on motivation
  Arms: Introductory PTSD module + TAU; Introductory PTSD module + one session of Shared Decision Making + individualised treatment
Behavioral: Shared Decision Making — A patient-centred shared decision making session where one of four standardised treatments can be chosen
  Arms: Introductory PTSD module + one session of Shared Decision Making + individualised treatment
Behavioral: Treatment as Usual — Treatment as usual
  Arms: Introductory PTSD module + TAU; Treatment as usual (TAU)
Behavioral: Standardised treatments — One of four treatments Treatment as ususal Sessions with psychologists Sessions with nurses Sessions with medical doctors
  Arms: Introductory PTSD module + one session of Shared Decision Making + individualised treatment

SUMMARY:
The goal of this clinical study is to improve the outcome of outpatient PTSD treatment at two clinics treating majority ethnic Danes and refugees with PTSD respectively. The study will consist of two similar randomized controlled trials.

The main questions the study aims to answer are:

* Does an added motivation enhancement module as a precursor for PTSD treatment reduce dropout and increase treatment outcome?
* Does an added Shared Decision-Making session which facilitate individualized treatment yield a superior outcome compared to PTSD treatment and PTSD treatment supplemented by motivation enhancement?

Participants are recruited at two different clinics, Psychotherapeutic Unit (PU) and Competence Centre for Transcultural Psychiatry (CTP). At PU the participants are randomized to one of two arms, and at CTP to one of three arms. One arm is the control group where participants will receive treatment as usual (TAU), one arm is the first intervention group where the participants will receive an Introductory PTSD module consisting of four sessions focusing on enhancing motivation for PTSD treatment, before continuing in TAU. The last arm is the second intervention group, which will only take place at CTP. Here the patient will receive the Introductory PTSD module followed by a session of Shared Decision Making, where the participant together with the MD decides which of four standardized treatment courses they will receive.

The treatment for all patients will last between 8-13 months.

DETAILED DESCRIPTION:
INTRODUCTION Traumatic events are a common experience worldwide. Data from the World Mental Health Consortium indicate that 70% of the general population reports at least one traumatic event, with 30.5% reporting four or more events. Certain populations, such as refugees and individuals in trauma-exposed professions (e.g., police officers, paramedics, and military personnel), are at heightened risk of encountering traumatic experiences. While the majority of individuals exposed to trauma do not develop long-term psychological distress, a significant subset develops posttraumatic stress disorder (PTSD), the primary mental health condition associated with trauma. According to the 2017 WHO World Mental Health Survey, 5.6% of trauma-exposed individuals develop PTSD, with half of these cases being persistent. PTSD is among the leading health-related causes of functional impairment, including days out of role.

Despite existing evidence-based interventions for PTSD, one-third of those undergoing treatment are non-responders and one-third drop out. This poses significant economic and social costs to the patient and to society. Previous randomized trials on refugees with PTSD at the CTP have pointed to motivation and cognitive resources as key predictors of treatment outcome. Others have theorized, and shown, that using standardized shared decision-making tools can enhance patient engagement in evidence-based PTSD treatment. Understanding the prerequisites of patients, such as motivational readiness and cognitive resources, are important in guiding decisions about treatment. At best, assigning homework or providing ambitious psychoeducation is a vain effort if the patient does not possess the motivation or cognitive means to engage, comply or fully understand. At worst, it demotivates and adds to the patient's sense of inadequacy.

These theories and hypotheses point to the need to gauge motivation, patient preference and values and assess cognition at the outset of treatment properly and to assess how to adapt treatment to fit each patient individually.

The overall aim of the PEP study is to improve the outcome of outpatient PTSD treatment.

1. To test the added value of the introductory PTSD module as a precursor of PTSD treatment in two RCTs. It is hypothesized that promoting patient engagement and motivation for treatment will increase treatment outcomes and reduce dropout relative to TAU.
2. To test the value of SDM to facilitate individualized treatment for the diverse population of refugees. This aim is specific to the CTP-trial. It is hypothesized that SDM + IPM will yield a superior outcome to TAU + IPM based on optimal utilization of resources of patients and clinicians.
3. To compare cognitive deficits in Danish civilians and trauma-affected refugees with PTSD, examining influences of emotional distress, demographic and socio-economic factors on test performance and to determine the predictive value of cognitive tests on treatment outcomes.
4. To study the association between motivation and severity of mental health symptoms, quality of life and functioning at baseline
5. To explore what patients and clinicians find useful and valuable about the introductory PTSD module add-on and SDM, and determine how these two components can influence treatment readiness and patient engagement
6. To examine the effect of treatment at six months follow-up on overall PTSD symptoms Course of treatment and data collection will follow the SPIRIT statement.

PATIENT RECRUITMENT Patients can be referred to the clinics by any MD, most often their general practitioner (GP), a private practicing psychiatrist or an MD from a mental health or somatic hospital. A senior psychiatrist at PU and CTP respectively assesses all referrals, and based on the referral, patients are invited for an initial assessment by a psychologist or MD at PU or an MD at CTP. At both clinics, if it is clear from the referral that the patient does not belong to the clinic's target group (i.e., does not present with trauma or any PTSD symptoms), the patient is not invited for an assessment.

Previous randomized trials at the CTP have included about 150 patients per year, and the fifth project) included 100 patients per year. The most recent study included 50 patients per year, but had significantly more restrictive inclusion criteria compared to the present study. In all trials 75-80 % of the patients have completed the project. No previous RCTs have been conducted at the PU, but it is estimated receiving 240 annual referrals for patients meeting the inclusion criteria.

Therefore, inclusion of 171 and 256 project participants, respectively, are deemed realistic within the given time frame.

INITIAL ASSESSMENT INITIAL ASSESSMENT AT PU The initial assessment is scheduled for all patients that are assessed to be in the target group as described above. The content of the assessment is not specific for this trial but applies to all initial assessments at PU, and no initiatives solely related to the trial will be performed during the initial assessment. The initial assessment at PU of the trauma-affected civilians is planned as 1-2 sessions (1-2 hours) and carried out by a member of the PTSD team. The team consists of authorized psychologists, unauthorized psychologists, psychologists with specialty in psychiatry and MDs. The assessment consists of a record of the trauma history, the main problem as seen by the patient, dispositions, social situation, somatic and psychiatric medical history, as well as a clinical and diagnostic assessment.

Standardized diagnostic tools such as part of Schedules for Clinical Assessment in Neuro-psychiatry (SCAN), International Trauma Interview (ITI) (80), and the ICD-10 research criteria will be applied in the interview. Various instruments of symptom severity and functioning are completed. After the initial assessment, the clinician presents the patient at a PTSD team conference. The team then collectively decides if the patient is eligible for treatment. To be eligible for treatment the patient must meet the criteria for PTSD and not have a psychotic disorder. The patient must be able to attend treatment, not be in current danger, and no longer be in the life situation that caused their PTSD. The patient should not be engaging in substance abuse or self-harm to a significant extent, and any other mental disorder must be well-managed enough for the patient to participate in trauma treatment.

Oral and written information about the treatment and the trial is given. If the patient fulfils eligibility criteria and consents to participate, the patient will be randomized after the initial assessment at PU.

INITIAL ASSESSMENT AT CTP The initial assessment is scheduled for all patients that are assessed to be in the target group of CTP as described above. The content of the assessment is not specific for this trial but applies to all initial assessments at CTP, and no initiatives solely related to the trial will be performed during the initial assessment. The initial assessment is planned as 2-4 sessions of approximately 45 minutes with an MD, resulting in a total of about two-three hours assessment and consists of: recording of the trauma history, the migration process, social situation, somatic and psychiatric medical history, as well as a clinical and diagnostic assessment. Standardized diagnostic tools such as part of Schedules for Clinical Assessment in Neuropsychiatry (SCAN), International Trauma Interview (ITI) (80), and the ICD-10 research criteria will be applied in the interview. Various instruments of symptom severity and functioning are completed.

Oral and written information about the treatment and the trial is given. If the patient fulfils eligibility criteria and consents to participate, the patient will be randomized after the initial assessment at CTP.

RANDOMISATION All patients will be randomized after a total of two to three-hour initial assessment with an MD or psychologist in accordance with inclusion and exclusion criteria. An equal number of patients are randomized into the trial arms of the two RCT's (total number of patients at PU is 171, and total number of patients at CTP is 256). The actual randomization is carried out in REDCap (Research Electronic Data Capture).

BLINDING Blinding patients and practitioners are not assessed to be appropriate due to the different nature of the treatment interventions. However, a blinded Hamilton (depression) rating, WHODAS 2.0 12-item, and WHODAS subscale on cognition will be carried out at the beginning and at the end of treatment. The group of raters, consisting of medical students, will be trained at CTP and will take part in regular joint ratings to ensure high quality and interrater reliability. Data assessment and data analysis will be performed blinded.

REPRESENTATIVITY Patients have not been selected based on more specific criteria than elsewhere in the treatment system and are therefore representative for the population at other clinics treating trauma-related mental health problems in an ethnic Danish and refugee population. The results can thus be generalized to other corresponding patient groups and are directly applicable in the planning of treatment for trauma-affected populations seeking outpatient treatment.

TRIAL FIDELITY To determine trial fidelity, patient attendance will be registered and after each consultation with a MD, psychologist, nurse or social counsellor, the topics addressed will be registered, as well as the methods used during the consultation and whether the patient has completed their exercises between sessions as planned. It will be registered whether the main content of the consultation was of social, psychological, or somatic character. At each consultation with an MD any changes in medication will also be recorded.

If patient IPM sessions or SDM session are cancelled a rescheduling will be attempted, but this may cause variation in timing of sessions in the treatment course. This will be registered. The use of the Problem Identification Form at sessions throughout the treatment is also registered.

VARIABILITY IN THE COURSE OF TREATMENT All patients will follow the treatment described above as accurate as possible, but due to the pragmatic nature of the study there will possibly be some variation in attendance and timing of meetings and sessions, as the patients may become ill or for some other reason do not show up for sessions or meetings.

FREQUENCY OF RATINGS Patients will be asked to complete self-ratings several times during treatment: at the diagnostic interview/assessment, and at the end of the treatment course. If more than one month passes between the diagnostic interview/assessment and the start of the IPM intervention or TAU for the control group, the patients will be asked to complete the self-ratings scales again. Furthermore, at 1) transition between IPM intervention and TAU/individualized treatment in the intervention groups or 2) after four sessions in the control groups the RPI will be completed.

Observer ratings including blinded Hamilton ratings will take place at the beginning and end of treatment, and PI administered at the first and fourth IPM session (intervention groups) or first and fourth session in TAU (control groups). Furthermore, at the beginning of TAU or the individualized treatment PGOMs will be completed.

In addition, some of the ratings will also be carried out at follow-up six months after end of treatment.

DATA COLLECTION Data will only be collected at PU and CTP. After each session the clinicians will fill out the case report form (CRF) in the research database through REDCap (Research Electronic Data Capture). All ratings will be carried out by a PU or CTP practitioner (MD, psychologist, nurse or social counsellor). Blinded observer-rated interviews of Hamilton D6, WHODAS 2.0 short version (level of cognition) and WHODAS 2.0 short version (level of functioning) will be carried out by medical students not linked to the team of practitioners, but to an independent rating team with thorough training in using the Hamilton rating scale and the WHODASs. To ensure quality and inter-rater reliability, the members in the rating team participate regularly in joint ratings under the guidance of one of the senior psychiatrists at CTP (six joint ratings per year). The investigators are overall responsible for the data collection.

DATA SECURITY All data collected for this project will be protected according to the General Data Protection Regulation (EU) 2016/679 (GDPR), the Danish Data Protection Act as well as the Danish Health Act. Information regarding the patients' health concerning history, the migration process, social situation, psychiatric medical history, medicine, allergies, abuse of drugs or alcohol and ratings will be passed on from the patient record to the investigators.

Data on somatic health issues are retrieved from Sundhedsplatformen during the period patients are receiving treatment at PU and CTP. Sociodemographic data are obtained from Statistics Denmark. These data extractions are detailed in the participant information provided with the consent for participation.

SOURCE DATA All data registered about the patients will be kept as source data in the form of original rating forms completed by the patients or practitioners, as well as structured patient records. Data will be saved for 15 years after the trial has ended, which will be stated in a letter of attorney signed by the patients. Case Report Form is source data, this will be described in the source data document, which will be filed in the Trial Master File.

QUALITY ASSURANCE Quality control and quality assurance will follow regular procedures as described in sections 3 and 4 of the Danish Executive Order on Good Clinical Practice (GCP). The first five RCTs at CTP have been under GCP monitoring, except the sixth and latest RCT, where the GCP unit had assessed that GCP monitoring was not necessary as CTP is assessed to have high-quality internal monitoring. This practice will be continued for the present study. The GCP unit has been contacted to inquire about the need for GCP monitoring for the present study.

The trials will be notified to the Danish Data Protection Agency (Datatilsynet) through the Capital Region of Denmark. Managing and filing data will be in accordance with current guidelines for research.

In order to ensure interrater reliability, all psychologists and MDs at PU and MDs at CTP will attend a SCAN course, all clinicians will attend a MI course, all MDs at CTP will attend a SDM course, and regular joint ratings including clinical assessment and observer-ratings will be carried out.

POWER CALCULATION The RCTs are powered individually and will be analyzed separately. Both trials are powered to detect a reduction in PTSD symptom scores equivalent to 0.5 standard deviation (SD) at a power level of 80% and a 5% significance level. A 0.5 SD reduction from baseline to end of treatment corresponds to a medium effect size and has been found to correspond well with the minimal clinically meaningful difference.

Previous studies have found ITQ standard deviations to vary across clinical PTSD populations but based on previous research and our own studies using the Harvard Trauma Questionnaire, it seems reasonable to expect that ½ SD will equal approximately 4 points on the ITQ. This is in line with what investigators consider the minimal clinically meaningful symptom reduction. This could, e.g., manifest as four symptoms decreasing in intensity from "extremely" to "quite a bit", or from "a little bit" to "not at all" from baseline to end of treatment.

At PU, which includes two randomized groups, these statistical assumptions result in a required completer sample of 64 participants per group, leading to a total of 128 completers.

The CTP RCT includes three randomized groups (two intervention groups and one treatment as usual [TAU] group), but will be powered to allow for pairwise comparisons between TAU and TAU + introductory PTSD module (IPM), as well as between IPM + TAU and IPM + shared decision making (SDM). This entails an identical power calculation to that of the PU RCT, resulting in a required completer sample of 64 participants per group. Across the three CTP groups, this leads to a required CTP completer sample of 192.

It is argued that the inclusion of SDM as a third arm in the CTP trial does not necessitate a correction for multiple testing because investigators evaluate distinct interventions rather than variations of a single treatment. This perspective is supported by Howard et al., who recommend that correction is only necessary when multiple hypotheses contribute to a single claim of effectiveness. Similarly, Wason et al. observed that correction for multiple testing in confirmatory multi-arm trials is most commonly applied in studies evaluating several doses or protocols of the same treatment.

In the CTP study, the hypotheses address distinct questions regarding the additive value of IPM to treatment-as-usual (TAU) and shared decision-making (SDM) as an alternative intervention. Because these hypotheses pertain to separate interventions, they do not constitute a "family" of hypotheses in the statistical sense. As such, the family-wise error rate (FWER) is not relevant, and no adjustment for multiple testing is necessary.

Correcting for an estimated 25% dropout, 171 participants will be included at PU, and 256 participants at CTP.

DROP-OUT ANALYSIS Drop-out analysis is based on the patients who show up at the pre-treatment assessment. The participants will be compared to the patients, who were excluded at the initial assessment on several dimensions in order to identify possible systematic selection bias. The participants included in the trials, but who eventually drop out and do not complete the trial, are included in the intention-to-treat analysis. In addition, completer analyses will be carried out.

DATA PROCESSING

1. The primary outcome variables are calculated as differences between baseline and end of treatment ratings. The differences between the two intervention groups at PU and the three intervention groups at CTP respectively can be measured with adjustment for baseline variables by ANCOVA and linear regression and with Full Information Maximum Likelihood (FIML) to handle missing data. All comparisons will be carried out separately for PU and CTP. In both cases, TAU will be compared to TAU + the motivational module. At the CTP, TAU + motivational module will additionally be compared to TAU + motivational module + shared decision making. If additional test proves relevant, these will be Bonferroni corrected for multiple testing.
2. Predictor analysis is carried out with regression models with outcome as dependent variable and patient characteristic as independent variable.
3. Cognitive test scores in the two samples will be assessed and compared. The factor structure of the test battery will be compared using confirmatory factor analysis. Hierarchical regression analyses will assess the influence of symptom severity and demographic variables on test scores, including acculturation in the CTP-sample. Additional analyses will investigate test-specific results and multiple regression analysis will be used to assess the relationship between cognitive test scores and treatment outcome.
4. Baseline: Different regression analyses will be applied to explore the relationship between motivation and severity of mental health symptoms, quality of life, and functioning.
5. Thematic qualitative analysis will be applied to explore what patients and clinicians find valuable about the IPM add-on and Shared Decision Making (SDM), and how these components influence treatment readiness and engagement.
6. Follow up outcome variables will be analyzed corresponding to 1.

Every session is registered during the trials to take account of the number of sessions in each group, when performing the analyses.

ELIGIBILITY:
In- and exclusion criteria of the randomised controlled trial for Psychotherapeutic Unit

Inclusion Criteria:

* Adults (18 years or older)
* PTSD pursuant to the ICD-10 research criteria
* Signed informed consent
* patients referred to "Main Level" treatment

Exclusion Criteria:

* Severe psychotic disorder (defined as patients with an ICD-10 diagnosis F2x and F30.1-F31.9). Participants are excluded only if the psychotic experiences are assessed to be part of an independent psychotic disorder and not part of a severe PTSD and/or depression.
* Dependence syndrome of drugs or alcohol: Active dependence and use (F1x.24-F1x.26).

In- and exclusion criteria of the randomised controlled trial for Competencecenter of Transcultural Psychiatry:

Inclusion criteria:

* Adult (18 years or older)
* Refugees or persons who have been family reunified with a refugee
* PTSD pursuant to the ICD-10 research criteria
* Psychological trauma experienced outside Denmark in the anamnesis. Trauma is imprisonment or detention with torture (according to the United Nations' definition of torture) or acts of cruel, inhuman and degrading treatment or punishment. Trauma can also be organised violence, long-term political persecution and harassment, or war and civil war experiences.
* Signed informed consent

Exclusion criteria:

* Severe psychotic disorder (defined as patients with an ICD-10 diagnosis F2x and F30.1-F31.9). Participants are excluded only if the psychotic experiences are assessed to be part of an independent psychotic disorder and not part of a severe PTSD and/or depression.
* Dependence syndrome of drugs or alcohol: Active dependence and use (F1x.24-F1x.26).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
International Trauma Questionnaire (ITQ) | Change from baseline to end-of-treatment after approximately 10 months
  A brief, simply worded measure, focusing only on the core features of PTSD and CPTSD, and employs straightforward diagnostic rules, based on the International Classification of Diseases, 11th edition (ICD-11). Scoring range: 0-4, lower scores reflect better outcome

SECONDARY OUTCOMES:
Readiness of Psychotherapy Index (RPI) | Change from baseline to after intervention after approximately 1,5 months
  RPI is used to assess an individual's readiness to engage in and benefit from psychotherapy. It evaluates motivation, perceived need for treatment, and confidence in the therapeutic process, helping clinicians gauge how prepared and willing a person is to start and actively participate in therapy. Scoring range: 1-5, in item 1, 2, 12, 13 and 17 a higher scores reflect lower degree of readiness, in item 3, 4, 5, 6, 7, 8, 9, 10, 11, 14, 15, 16, 18, 19 og 20 a higher score reflects a higher degree of readiness
Hopkins Symptom Check List-25 (HSCL) | Change from baseline to end-of-treatment after approximately 10 months
  HSCL-25 is an internationally applied and thoroughly validated self-administered rating scale assessing the severity of anxiety and depression symptoms. This is a short version of the Symptom Checklist-90 (SCL-90). It consists of 25 questions, 10 regarding anxiety and 15 regarding depression. Scoring range: 1-4, lower scores reflect better outcome
Psychological Outcome Profiles questionnaire (PSYCHLOPS) | Change from baseline to end-of-treatment after approximately 10 months
  It is a self-report measure designed to assess patient-generated outcomes measuring three domains: Problems, Function and Wellbeing.
  There is a pre-treatment and a post-treatment version. Scoring range: 0-5, lower score reflect better outcome
World Health Organisation - 5 Well-being Index (WHO-5) | Change from baseline to end-of-treatment after approximately 10 months
  It is a self-administered questionnaire evaluating quality of life, consisting of five questions with each six possible answers. The questionnaire has been used to assess the quality of life in several psychiatric diagnostic groups. In addition, the scale has been used to assess overall treatment effects in the field of psychiatry. Scoring range: 0-100, higher scores reflect better outcome.
Life Events Checklist for DSM-5 (LEC-5) | Administered once at the initial assessment
  The Life Events Checklist for DSM-5 (LEC-5) is a self-report measure developed to find potentially traumatic events in a patient's lifetime. The LEC-5 assesses exposure to 16 potentially traumatic events and includes an additional item for any other extraordinarily stressful events.
Post-migration Living Difficulties Check List (PMLD) | Administered once at the initial assessment, but only at CTP
  It is a self-administered rating scale examining the extent to which post-migration challenges has been a problem for the patient, originally over the past 12 months. Scoring range: 0-68, lower scores reflect better outcome.
The 9-item Shared Decision Making questionnaire (SDM-Q-9) | Administered once during treatment at the shared decision-making session only at CTP
  It assesses the extent of collaboration in healthcare decision-making. It ensures patient preferences are integrated into clinical decisions, enhancing patient-centred care and communication, leading to better health outcomes and satisfaction. Scoring range: 1-6, higher scores reflect better outcome.
The World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Change from baseline to end-of-treatment after approximately 10 months
  the interviewer administered 12-item short version, is an observer rating scale used to measure health and disability across cultures in six core life domains of cognition/communication, mobility, self-care, interpersonal interaction, life activities, and participation in society. The items are rated on a 5-point Likert scale of functional impairment (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). The WHODAS has been widely used across epidemiological surveys worldwide proving sound internal consistency (Cronbach α=0.87 for the entire scale) and test-retest reliability (intraclass correlation coefficients ranging from 0.69 to 0.89 across items).
The World Health Organization Disability Assessment Schedule (WHODAS 2.0), cognition | Change from baseline to end-of-treatment after approximately 10 months
  A subscale on cognition is an observer rating scale with 6 questions used to assess concentration, memory, problem solving, learning and communication. Scoring range: 0-30, lower scores reflect better outcome.
Hamilton depression scale (HAM-D6) | Change from baseline to end-of-treatment after approximately 10 months
  It is an observer rating scale assessing depression on the basis of semi-structured interviews. The scales have been used widely in psychiatric research including on trauma-affected refugees. Scoring range: 0-22, lower scores reflect better outcome.
Global Assessment of Functioning - Symptoms (GAF-S) | Time Frame: Change from baseline to end-of-treatment after approximately 10 months
  Observer rating scale used to assess the degree of symptoms. Scoring range: 1-100, higher scores reflect better outcome. Scoring range: 1-100, higher scores reflect better outcome.
Global Assessment of Functioning - Functioning (GAF-F) | Change from baseline to end-of-treatment after approximately 10 months
  Observer rating scale used to assess the degree of social and psychological functioning. Scoring range: 1-100, higher scores reflect better outcome.
Shared Decision Making questionnaire - physician version (SDM-Q-Doc) | Administered once during treatment at the shared decision-making session only at CTP
  It is an adapted version of the SDM-Q-9, which measures the degree of patient involvement in a physician consultation from the perspective of the physician. Scoring range: 1-6, higher scores reflect better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Carlsson, Study Chair — Mental Health Services in th Capital Region, Denmark
Locations (1):
- Mental Health Centre Ballerup, Ballerup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No